CLINICAL TRIAL: NCT05264441
Title: Choice of Inhalation Device in Asthma and COPD Patients
Brief Title: Choice of Inhalation Device
Acronym: Choice Device
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Choice Device
Record Dates: First submitted 2022-02-04; First posted 2022-03-03 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2021-09

CONDITIONS: Asthma; COPD
Keywords: Inhaler Device; In-Check DIAL G16
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Cross sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Asthma and COPD patients (Other): There will be only 1 arm in this study. COPD and asthma patients will be in the same arm.
  Interventions: Device: In-Check DIAL G16

INTERVENTIONS:
Device: In-Check DIAL G16 — Patients will inspire into an In-Check DIAL G16 device.

SUMMARY:
In this study, asthma and COPD patients will be invited to participate after the consultation with their pulmonologist.

The intervention consists of three steps. The first step is to perform a deep inspiration. The second step is to demonstrate the correct use of a pMDI. The third step is to perform a strong inspiration into the In-Check Dial device over 5 different resistances.

DETAILED DESCRIPTION:
The study will take place in the respiratory outpatient clinic. Patients will be invited to participate in the study after the consultation with the pulmonologist. All pulmonologists have a flowchart regarding the optimal choice of inhaler at their disposition.

Patients will be provided sufficient time to read the informed consent file and to ask questions about the study. After giving their informed consent they will be screened for eligibility by an investigator. Demographic data and characteristics will be retrieved from the medical record (EMD) of study participants.

The intervention will consist of three different steps.

First, the patient will perform a deep voluntary inspiration. The patient's ability to perform this inspiration will be assessed and scored by the investigator.

Secondly, the peak inspiratory flows (PIF) will be measured with an In-check Dial device over 5 different resistances.

The minimal and optimal peak inspiratory flow rates (PIFRs) differ by device. A minimum flow of 30 L/min is required for most DPI's. The optimal flow varies from 30 L/min to 35, 45, 50, 60 or 65 L/min.

Due to the fact that there is still discussion about the effectiveness of PIF's going from 30 to 60 L/min, an arbitrary cut-off value will be set at 45 L/min. This cut-off value for sufficient PIF will be measured over a moderate resistance to distinguish subtherapeutic from therapeutic levels. If the patient reaches a PIF lower than 45 L/min, the patient will be asked to make a second attempt.

Subsequently, the patient will receive education about the correct coordination, which is necessary in the use of dose inhalers. The patient will be evaluated for sufficient actuation-inhalation coordination, through a placebo pMDI.

The evaluation of the voluntary deep inspiration, PIF and coordination will be by pass or fail evaluation. Subsequently, the fitness of a patient to use any of the three inhaler classes will be determined by using a diagram designed by a Belgian expert group (unpublished to date; courtesy of Didier Cataldo, ULiège).

If a mismatch between prescribed inhaler and suitable inhaler types is found, the treating physician of the patient will be informed. By doing so, the investigators wish to avoid patients receiving prescriptions for inhalers that they cannot use properly.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients (GOLD II-IV)
* Patients with severe asthma
* Patients with mild-to moderate asthma aged < 70y
* Patients with asthma aged ≥ 70y

Exclusion Criteria:

* Patients with asthma or COPD not on inhaled therapy for maintenance treatment
* Patients younger than 18y
* Patients unable to give their informed consent due to mental or physical disability
* Patients who don't speak French or Dutch

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with device mismatch | up to 2 months
  Data from COPD and asthma patients will be compared

DOCUMENTS (1):
  • Study Protocol (2021-03-05): https://cdn.clinicaltrials.gov/large-docs/41/NCT05264441/Prot_000.pdf